CLINICAL TRIAL: NCT01457092
Title: Self-expandable, Fully Covered Metal Stents in Biliary Strictures Due to Chronic Pancreatitis Not Responding to Plastic Stenting: a Prospective Study With Two Years Follow-up.
Brief Title: Self-expandable, Fully Covered Metal Stents in Biliary Strictures Due to Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Guido Costamagna, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A/1530/2005
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Benign Biliary Strictures; Chronic Pancreatitis
Keywords: benign biliary strictures; chronic pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FC Nitinol SEMS (Experimental): FC Nitinol SEMS
  Interventions: Device: FC Nitinol SEMS (Niti-S, TaeWoong Medical Co., Korea)

INTERVENTIONS:
Device: FC Nitinol SEMS (Niti-S, TaeWoong Medical Co., Korea) — Placement of self-expandable metal stents

SUMMARY:
The purpose of the study was to analyze the resolution rate of benign biliary strictures due to chronic pancreatitis after temporary insertion of unflared-ends and flared-ends fully covered self-expandable metal stents.

DETAILED DESCRIPTION:
Endoscopic treatment of benign biliary strictures include the placement of plastic stents or Self-Expandable Metal Stents. Long term results of placement of a single plastic stent are disappointing. Better results have been obtained by endoscopic insertion of multiple plastic stents.

Biliary Self-Expandable Metal Stents used for malignant strictures are uncovered or partially covered with a plastic coating. More recently, fully covered SEMS have been developed and are now available on the market and due to their removability are proposed also for benign indications.

Uncovered and partially covered biliary Self-Expandable Metal Stents for chronic pancreatitis-related benign biliary strictures on long-term may clog due to tissue ingrowth through the uncovered meshes.

Removable fully covered Self-Expandable Metal Stents seem to be an attractive option for CP-related BBS, but scarce data are available in the literature.

The investigators conducted a feasibility, prospective, tertiary single-centre trial to investigate the durable resolution of chronic pancreatitis-related benign biliary strictures after temporary insertion of FC SEMS with unflared-ends and flared-ends.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years,
2. symptomatic (persistent cholestasis, jaundice, cholangitis) common bile duct strictures secondary to CP, that persist 3 months or more after placement of a single 10 French plastic stent and
3. patient unfit for surgery (portal cavernomatosis, comorbidities) or patient refusal of surgery.

Exclusion Criteria:

1. benign biliary strictures secondary to compression from a pancreatic pseudocyst;
2. patients with associated pancreatic neoplasia
3. ongoing alcohol abuse (ethanol > 80 g/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Stricture dilatation | 6 months